CLINICAL TRIAL: NCT03927144
Title: A 12-month Prospective, Randomized, Interventional, Global, Multi-center, Active-controlled Study Comparing Sustained Benefit of Two Treatment Paradigms (AMG334 qm vs. Oral Prophylactics) in Adult Episodic Migraine Patients
Brief Title: Study of Sustained Benefit of AMG334 in Adult Episodic Migraine Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMG334A2401; 2018-001228-20 (EudraCT Number); CAMG334A2401 (Other: Novartis)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Episodic Migraine
Keywords: Erenumab; AMG334; Migraine; Episodic; Headache; CGRP
MeSH Terms: conditions — Migraine Disorders; Recurrence; Headache | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMG334 70 mg/140 mg (Experimental): Participants were randomized to receive 70 mg or 140 mg of AMG334 as a subcutaneous injection once per month for 52 weeks in the Core Phase.
  Participants were permitted to switch to an approved oral prophylactic based on treatment failure status and at the investigator's and participant's discretion.
  Participants who completed visits through Week 52 of the Core Phase were eligible to participate in the 52-week Extension Phase of the study.
  Interventions: Drug: AMG334; Drug: Oral Prophylactic
- Oral Prophylactic (Active Comparator): Participants were randomized to receive a standard of care (SOC) locally approved oral prophylactic migraine medication once per day for 52 weeks in the Core Phase, as prescribed per local country labels.
  Participants were permitted to switch to a different approved oral prophylactic based on treatment failure status and at the investigator's and participant's discretion.
  Participants who completed visits through Week 52 of the Core Phase were eligible to participate in the 52-week Extension Phase of the study.
  Interventions: Drug: AMG334; Drug: Oral Prophylactic

INTERVENTIONS:
Drug: AMG334 — Subcutaneous Injection
  Other Names: Erenumab
Drug: Oral Prophylactic — SOC Oral Tablet/Capsule

SUMMARY:
The purpose of this study is to compare the sustained long-term benefit between two treatment paradigms of migraine prophylactic agents (erenumab versus a control arm of oral prophylactics) in episodic migraine patients who have previously failed 1 to 2 prophylactic migraine treatments.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Adults greater than or equal to 18 years of age upon entry into screening.
* Documented history of migraine (with or without aura) greater than or equal to 12 months prior to screening according to the International Classification of Headache Disorders-3rd Edition (ICHD-3).
* Greater than or equal to 4 and less than 15 days per month of migraine symptoms (based on ICHD-3 criteria) on average across 3 months prior to screening based on retrospective reporting.
* Less than 15 days per month of headache symptoms (i.e., migraine and non-migraine).
* Subjects in need for switching by documented failure of 1 or 2 prophylactic treatments in the last 6 months due to either lack of efficacy or poor tolerability. For subjects with 1 prior treatment failure, the failure should have occurred in the last 6 months. For subjects with 2 prior treatment failures, the second treatment failure should have occurred in the last 6 months.
* During baseline: Confirmed migraine frequency of 4 to 14 migraine days and less than 15 days of headache symptoms.
* During baseline: greater than or equal to 80% compliance with the headache diary.

Exclusion Criteria:

* Subjects meeting any of the following criteria are not eligible for inclusion in this study.

  * Older than 50 years of age at migraine onset.
  * History of cluster headache or hemiplegic migraine headache.
  * Unable to differentiate migraine from other headaches.
  * Lack of efficacy or poor tolerability with greater than 2 treatments from the 7 medication categories for prophylactic treatment of migraine after an adequate therapeutic trial.
* Efficacy failure is defined as no meaningful reduction in headache frequency, duration, and/or severity after administration of the medication for at least 6 weeks at the generally accepted therapeutic dose(s) based on the investigator's assessment.
* Tolerability failure is defined as documented discontinuation due to adverse events of the respective medication during the last 6 months prior to screening.
* The following scenarios do not constitute lack of therapeutic response:
* Lack of sustained response to a medication.
* Patient decision to halt treatment due to improvement.
* Used a prohibited medication from the 7 categories of prior prophylactic medications within 3 months prior to the start of and during baseline for a non-migraine indication if dose is not stable
* Exposure to botulinum toxin in the head and/or neck region within 4 months.
* Taken the following for any indication in any month during the 2 months prior to the start of the baseline period:

  * Ergotamines or triptans on greater than or equal to 10 days per month, or Simple analgesics (non-steroidal anti-inflammatory drugs [NSAIDs], acetaminophen) on greater than or equal to 15 days per month, or
  * Opioid- or butalbital-containing analgesics on greater than or equal to 4 days per month.
* Device, or procedure that potentially may interfere with the intensity or number of migraine days within 2 months prior to the start of or during baseline.
* History of major psychiatric disorders (such as schizophrenia or bipolar disorder) or current evidence of depression. Subjects with anxiety disorder and/or major depressive disorders are permitted in the study if they are considered by the investigator to be stable and are taking no more than 1 medication for each disorder. Subjects must have been on a stable dose within the 3 months prior to the start of the baseline period.
* History of seizure disorder or other significant neurological conditions other than migraine. Note: a single childhood febrile seizure is not exclusionary.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Human immunodeficiency virus (HIV) infection by history.
* History or evidence of any other unstable or clinically significant medical condition or clinically significant vital sign, laboratory, or electrocardiogram (ECG) abnormality during that could pose a risk to subject safety or interfere with the study evaluation.
* Myocardial infarction, stroke, transient ischemic attack, unstable angina, or coronary artery bypass surgery or other re-vascularization procedures within 6 months prior to screening.
* Score "yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS, if this ideation occurred in the past 6 months, or "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self-Injurious Behavior" (item also included in the Suicidal Behavior section), if this behavior occurred in the past 2 years.
* Evidence of drug or alcohol abuse or dependence, based on Investigator discretion within 12 months.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential must use contraception during dosing with study treatment.
* Use of other investigational drugs within 5 half-lives of enrollment, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
* History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes.
* Previous exposure to AMG334 or exposure to any other prophylactic CGRP-targeted therapy (prior to the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (112):
- United States (20):
  - Stanford Headache Center, Stanford, California
  - Yale Center for Clinical Research, New Haven, Connecticut
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - George Washington Hospital, Washington D.C., District of Columbia
  - University of Miami Headache Division, Miami, Florida
  - Premier Research Institute, West Palm Beach, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - Robbins Headache Clinic, Riverwoods, Illinois
  - Medvadis, Watertown, Massachusetts
  - New England Regional Headache Center, Inc, Worcester, Massachusetts
  - MHNI, Ann Arbor, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Headache Center, Ridgeland, Mississippi
  - Study Metrix Research, City of Saint Peters, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Laszlo Mechtler, Amherst, New York
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Texas Neurology, Dallas, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
- Argentina (3):
  - IDIM Instituto de Investigaciones Metabolicas, Buenos Aires
  - Mautalen Salud e Investigacion, Ciudad Autonoma de Bs As
  - Centro Medico Privado en Reumatologia, San Miguel de Tucumán
- Austria (3):
  - Univ. Klinik fuer Neurologie, Innsbruck
  - Ordensklinikum Linz Barmherzigen Schwestern, Linz
  - Univ Klinik fuer AKH, Vienna
- Belgium (6):
  - AZ Sint Jan, Bruges
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - Jessa Ziekenhuis- Campus Virga Jesse Dienst Gastro-entrologie, Hasselt
  - Heilig Hart Ziekenhuis Lier, Lier
  - Centre Hospitalier Regional de la Citadelle, Liège
- Czechia (9):
  - Neurologicka ambulance Quattromedica, Brno
  - NEUROHK sro, Choceň
  - Brain Soultherapy sro, Kladno
  - DADO Medical S R O, Prague
  - Thomayerova Nemocnice, Prague
  - Forbeli SRO, Prague
  - Institut neuropsychiatricke pece, Prague
  - Clintrial SRO, Prague
  - Vestra Clinics sro, Rychnov nad Kněžnou
- Finland (3):
  - Terveystalo Ruoholahti, Helsinki
  - Laakarikeskus Aava Itakeskus, Helsinki
  - Terveystalo Pulssi, Turku
- France (5):
  - CHRU de LILLE, Lille
  - Hopital Lariboisiere Centre d Urgence des Cephalees, Paris
  - Hopital Charles Nicolle Departement de Neurologie, Rouen
  - CH Yves Le Foll, Saint-Brieuc
  - CHU St Etienne Hopital Nord Bat A, Saint-Etienne
- Germany (5):
  - GP Dept of Neurology, Bochum
  - Neurologische Gemeinschaftspraxis Klemt & Bauersachs, Dortmund
  - Neurologische Gemeinschaftpraxis im Bienenkorbhaus, Frankfurt
  - AmBeNet Hausarztpraxis, Leipzig
  - Medamed GmbH Studienambulanz, Leipzig
- Greece (7):
  - Navy Hospital of Athens "NNA" Main Centre, Athens
  - Aeginition Hospital of Athens, University of Athens, Athens
  - Neurologicka Ambulancia Konzilium s r o, Athens
  - 401 Army General Hospital of Athens Main Centre, Athens
  - MEDITERRANEO Hospital, Glyfada
  - General Hospital of Patra O AGIOS ANDREAS Neurology Clinic, Pátrai
  - Euromedica General Clinic of Thessaloniki Neurology Dept, Thessaloniki
- Ireland (2):
  - Bon Secours Hospital, Cork
  - Beaumont Hospital, Dublin
- Israel (5):
  - Hillel Yaffe MC, Hadera
  - Rambam Medical Center, Haifa
  - Laniado, Netanya
  - Sheba MC, Ramat Gan
  - Tel Aviv Sourasky Medical Center Ichilov, Tel Aviv
- Italy (6):
  - A O Perugia Osp S Maria Misericordia Loc S Andrea d Fratte, Perugia, PG
  - IRCCS San Raffaele Pisana, Roma, RM
  - Ospedali Riuniti Torrette di Ancona, Ancona
  - ASST degli Spedali Civili di Brescia Univ degli Studi, Brescia
  - Policl.Universit.Campus Bio-Medico Università Campus Bio-Med U.O.C.Area di Oncologia Medica, Roma
  - Azienda Ospedaliera Sant'Andrea - Università La Sapienza, Roma
- Netherlands (4):
  - Zuyderland Medisch Centrum, Geleen
  - Martini Ziekenhuis, Groningen
  - Canisius Wilhelmina Hospital Dept of Neurology C-70, Nijmegen
  - Isala Ziekenhuis, Zwolle
- Poland (5):
  - Centrum Leczenia Padaczki i Migreny, Krakow
  - Gabient Lekarski Jacek Rozniecki, Lodz
  - OHA MED Sp zo o, Warsaw
  - ETG Warszawa, Warsaw
  - Wojskowy Instutyt Medyczny CSK MON, Warsaw
- Portugal (5):
  - Hospital Garcia de Orta EPE, Almada
  - Hospital da Luz, Lisbon
  - Hospital Santa Maria, Lisbon
  - Hospital Pedro Hispano Matosinhos E P E, Matosinhos Municipality
  - Centro Hospitalar do Porto Hospital Geral de Santo Antonio Serviço de Neurologia, Porto
- Slovakia (6):
  - MUDr Beata Dupejova s r o, Banská Bystrica
  - Nemocnica sv Michala a s, Bratislava
  - Nemocnica Komarno s r o, Komárno
  - Neurologicke oddelenie VNsP Levoca, Levoča
  - Neurolog odd NsP Liptovsky Mikulas, Liptovský Mikuláš
  - Neurologicka a algeziologicka ambulancia SANERA s r o, Prešov
- Spain (9):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Clinico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Vall D'Hebron, Barcelona, Catalonia
  - Hospital Clinico Universitario Valencia, Valencia, Communidad Valencia
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital La Paz, Madrid
  - Hospital Marques de Valdecilla, Santander
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- United Kingdom (9):
  - Queen Elizabeth Hospital Pharmacy Dept., Edgbaston, Birmingham
  - The John Radcliffe Hospital, Headington, Oxfordshire
  - University Hospital of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire
  - Glasgow Clinical Research Facility, Glasgow
  - Hull and amp East Yorkshire Hospitals NHS Trust, Hull
  - St Thomas Hospital, London
  - King's College Hospital London, London
  - Royal Victoria Infirmary, Newcastile Upon Tyne
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No
Data sharing for this study is the responsibility of Novartis. Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Pozo-Rosich P, Dolezil D, Paemeleire K, Stepien A, Stude P, Snellman J, Arkuszewski M, Stites T, Ritter S, Lopez Lopez C, Maca J, Ferraris M, Gil-Gouveia R. Early Use of Erenumab vs Nonspecific Oral Migraine Preventives: The APPRAISE Randomized Clinical Trial. JAMA Neurol. 2024 May 1;81(5):461-470. doi: 10.1001/jamaneurol.2024.0368. PMID 38526461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 621 participants were enrolled at 84 centers in Argentina, Austria, Belgium, Czechia, Finland, France, Germany, Greece, Israel, Italy, the Netherlands, Poland, Portugal, Slovakia, Spain, the United Kingdom and the United States.
  The primary completion date based on the Core Phase was 01-Oct-2021. The study completion date was 30-Sep-2022.
Pre-assignment Details: Participants were randomized 2:1 [AMG334 70/140 mg: oral prophylactic].
  Randomization was stratified by prior prophylactic migraine medication treatment failure (due to insufficient efficacy or poor tolerability) reported during Screening/Baseline Period: 1 treatment failure (TF1) vs 2 treatment failures (TF2). A 30% cap of randomized participants to the TF2 strata was implemented. The stratification and 30% cap were implemented within Interactive Response Technology.
Groups:
- AMG334 70 mg/140 mg: Participants received 70 mg or 140 mg of AMG334 as a subcutaneous injection once per month for 52 weeks in the Core Phase.
  Participants were permitted to switch to an approved oral prophylactic based on treatment failure status and at the investigator's and participant's discretion.
  Eligible Core Phase completers (completed Week 52 and were benefitting from AMG334 treatment) entered the Extension Phase to continue to receive 70 mg or 140 mg AMG334 for up to 52 weeks.
- Oral Prophylactic: Participants received a standard of care (SOC) approved oral prophylactic once per day for 52 weeks in the Core Phase, as prescribed per local country labels.
  Participants were permitted to switch to a different approved oral prophylactic based on treatment failure status and at the investigator's and participant's discretion.
  Eligible Core Phase completers (completed Week 52 and were in need of a treatment switch) entered the Extension Phase to receive 70 mg or 140 mg AMG334 for up to 52 weeks.
Period: Core Phase
Arm/Group | AMG334 70 mg/140 mg | Oral Prophylactic
Started | 413 | 208
Completed (Completed 52 week core phase) | 377 | 146
Not Completed | 36 | 62
Not completed — Adverse Event | 9 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — New Therapy for Study Indication | 0 | 1
Not completed — No Longer Clinically Benefiting | 4 | 4
Not completed — Physician Decision | 2 | 8
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 16 | 40
Period: Extension Phase
Arm/Group | AMG334 70 mg/140 mg | Oral Prophylactic
Started | 343 (Eligible core phase completers (completed Week 52 and were benefitting from AMG334 treatment) entered the extension phase) | 118 (Eligible core phase completers (completed Week 52 and were in need of a treatment switch) entered the extension phase)
Completed | 328 | 108
Not Completed | 15 | 10
Not completed — Adverse Event | 2 | 1
Not completed — No longer clinically benefiting | 4 | 5
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 8 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): Included all participants to whom study treatment had been assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG334 70 mg/140 mg | Oral Prophylactic | Total
Number analyzed (Participants) | 413 | 208 | 621
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11.5) | 41.5 (10.4) | 41.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 363 | 182 | 545
  Male | 50 | 26 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 406 | 206 | 612
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 17 | 42
  Not Hispanic or Latino | 381 | 190 | 571
  Not Reported | 6 | 1 | 7
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Initially Assigned Treatment and Achieved at Least a 50% Reduction From Baseline in Monthly Migraine Days at Month 12
Description: A migraine day was defined as any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine with or without aura, lasting for ≥ 30 minutes, and meeting at least one of the following criteria:
  1. ≥2 of the following pain features:
     * Unilateral
     * Throbbing
     * Moderate to severe
     * Exacerbated with exercise/physical activity
  2. ≥1 of the following associated symptoms:
     * Nausea and/or vomiting
     * Photophobia and phonophobia
  If the participant took a migraine-specific medication (ie, triptan or ergotamine) during aura, or to treat a headache on a calendar day, then it was counted as a migraine day regardless of the duration and pain features/associated symptoms.
  In addition to achieving at least a 50% reduction from baseline in monthly migraine days, participants must have also completed their initially assigned treatment through Month 12.
Time Frame: Baseline and Month 12
Population: FAS: Included all participants to whom study treatment had been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG334 70 mg/140 mg | Oral Prophylactic
Number analyzed (Participants) | 413 | 208
Participants | 232 | 35
Statistical Analysis 1: Comparison: AMG334 70 mg/140 mg vs Oral Prophylactic; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted for stratification factor (no. of prior prophylactic migraine treatment failures=1 vs 2) after missing data were imputed as non-response; Odds Ratio (OR) = 6.48, 95% CI 2-sided [4.28 to 9.82]

2. Secondary Outcome: Number of Participants Who Completed Initially Assigned Treatment at Month 12
Time Frame: Month 12
Population: FAS: Included all participants to whom study treatment has been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG334 70 mg/140 mg | Oral Prophylactic
Number analyzed (Participants) | 413 | 208
Participants | 359 | 78
Statistical Analysis 1: Comparison: AMG334 70 mg/140 mg vs Oral Prophylactic; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted for number of prior prophylactic migraine treatment failures=1 vs 2 after missing data were imputed as non-response; Odds Ratio (OR) = 11.27, 95% CI 2-sided [7.53 to 16.87]

3. Secondary Outcome: Cumulative Mean Change From Baseline on the Monthly Migraine Days to Week 52
Description: A migraine day was defined as any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). The mean of monthly migraine days was obtained cumulatively every 4 weeks across 52 weeks (for example, at Week 8 the mean will be based on data from Week 1 to Week 8; and at Week 12 the mean will be based on data from Week 1 to Week 12). The cumulative mean change from baseline in monthly migraine days was derived using difference between cumulative average of each month and baseline monthly migraine days.
Time Frame: Baseline and Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, and Week 52
Population: Participants in the FAS with data available at each time point. The FAS included all participants to whom study treatment had been assigned. All participants included in the overall number of participants analyzed contributed to the post-baseline data for this endpoint.
Measure: Mean (Standard Error); unit: migraine days per month
Arm/Group | AMG334 70 mg/140 mg | Oral Prophylactic
Number analyzed (Participants) | 413 | 208
migraine days per month
  Week 4: number analyzed (Participants) | 406 | 184
  Week 4 | -2.55 (0.17) | -0.55 (0.25)
  Week 8: number analyzed (Participants) | 404 | 151
  Week 8 | -3.00 (0.17) | -1.01 (0.25)
  Week 12: number analyzed (Participants) | 399 | 131
  Week 12 | -3.27 (0.17) | -1.05 (0.26)
  Week 16: number analyzed (Participants) | 398 | 121
  Week 16 | -3.45 (0.17) | -1.22 (0.26)
  Week 20: number analyzed (Participants) | 391 | 111
  Week 20 | -3.63 (0.17) | -1.35 (0.26)
  Week 24: number analyzed (Participants) | 387 | 101
  Week 24 | -3.75 (0.17) | -1.56 (0.26)
  Week 28: number analyzed (Participants) | 383 | 94
  Week 28 | -3.84 (0.17) | -1.73 (0.26)
  Week 32: number analyzed (Participants) | 378 | 89
  Week 32 | -3.93 (0.17) | -1.91 (0.27)
  Week 36: number analyzed (Participants) | 375 | 83
  Week 36 | -3.99 (0.17) | -1.99 (0.27)
  Week 40: number analyzed (Participants) | 371 | 82
  Week 40 | -4.05 (0.17) | -2.06 (0.27)
  Week 44: number analyzed (Participants) | 368 | 80
  Week 44 | -4.12 (0.17) | -2.11 (0.27)
  Week 48: number analyzed (Participants) | 365 | 78
  Week 48 | -4.18 (0.17) | -2.07 (0.27)
  Week 52: number analyzed (Participants) | 359 | 78
  Week 52 | -4.24 (0.17) | -2.11 (0.27)
Statistical Analysis 1: Comparison: AMG334 70 mg/140 mg vs Oral Prophylactic; Comparison of mean change from baseline in monthly migraine days at Week 52; Test type: Superiority; p < 0.001, Linear mixed effects model; Treatment difference = -2.13, 95% CI 2-sided [-2.74 to -1.52], Standard Error of Mean 0.31 — AMG334 70 mg/140 mg vs Oral Prophylactic

4. Secondary Outcome: Number of Responders as Measured by the Patient's Global Impression of Change (PGIC) Scale at Week 52
Description: The PGIC scale consists of one item which measures the participants' perception of change in their condition relative to the beginning of the study. Responses are rated on a 7-item response scale ranging from very much improved (7) to no change or worsened condition (1). A responder was defined as a participant with a PGIC score of at least 5 (5=moderately better, 6=better, 7=a great deal better), at Week 52 for participants who completed the treatment period at Week 52 on the initially assigned treatment.
Time Frame: Baseline and Week 52
Population: FAS: Included all participants to whom study treatment had been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG334 70 mg/140 mg | Oral Prophylactic
Number analyzed (Participants) | 413 | 208
Participants | 314 | 39
Statistical Analysis 1: Comparison: AMG334 70 mg/140 mg vs Oral Prophylactic; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 13.75, 95% CI 2-sided [9.08 to 20.83]

ADVERSE EVENTS:
Time Frame: Day 1 to Week 52 of the Core Phase and Day 1 to Week 52 of the Extension Phase
Description: An adverse event (AE) was defined as any untoward medical occurrence (e.g., any unfavorable & unintended sign [including abnormal laboratory findings], symptom or disease) in a participant after the first dose of study treatment.
  AEs were collected based on treatment type received (AMG334 versus oral prophylactic) and were not collected separately for each dose.
  The Safety Set: Included all participants who received at least one dose of study treatment.
Groups:
- Core Phase: AMG334 70mg/140mg: Participants received 70 mg or 140 mg of AMG334 as a subcutaneous injection once per month for 52 weeks in the Core Phase. Participants were permitted to switch to an approved oral prophylactic based on treatment failure status and at the investigator's and participant's discretion.
  Includes 9 participants who switched from AMG334 to SOC oral prophylactics during the core phase; only AEs prior to the treatment switch to SOC oral prophylactics are reported.
- Core Phase: Oral Prophylactics: Participants received a SOC approved oral prophylactic once per day for 52 weeks in the Core Phase, as prescribed per local country labels. Participants were permitted to switch to a different approved oral prophylactic based on treatment failure status and at the investigator's and participant's discretion.
  Includes 9 participants who switched from AMG334 to SOC oral prophylactics during the core phase; only AEs following the treatment switch to SOC oral prophylactics are reported.
- Extension Phase: AMG334 70mg/140mg Continuing on AMG334 70mg/140mg: Eligible Core Phase completers (completed Week 52 and were benefitting from AMG334 treatment) entered the Extension Phase to continue to receive 70 mg or 140 mg AMG334 for up to 52 weeks.
- Extension Phase: Oral Prophylactics Then AMG334 70mg/140mg: Eligible Core Phase completers (completed Week 52 and were in need of a treatment switch) who received a SOC approved oral prophylactic in the Core Phase entered the Extension Phase to receive 70 mg or 140 mg AMG334 for up to 52 weeks.
Arm/Group | Core Phase: AMG334 70mg/140mg | Core Phase: Oral Prophylactics | Extension Phase: AMG334 70mg/140mg Continuing on AMG334 70mg/140mg | Extension Phase: Oral Prophylactics Then AMG334 70mg/140mg
All-Cause Mortality (participants affected / at risk) | 0/408 | 0/206 | 0/343 | 0/118
Serious Adverse Events (participants affected / at risk) | 15/408 | 9/206 | 9/343 | 4/118
Other Adverse Events (participants affected / at risk) | 131/408 | 91/206 | 106/343 | 47/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Phase: AMG334 70mg/140mg (N=408) | Core Phase: Oral Prophylactics (N=206) | Extension Phase: AMG334 70mg/140mg Continuing on AMG334 70mg/140mg (N=343) | Extension Phase: Oral Prophylactics Then AMG334 70mg/140mg (N=118)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Medical device pain (General disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureteric rupture (Renal and urinary disorders) | 0 | 0 | 1 | 0
Breast fibrosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Skin laxity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Phase: AMG334 70mg/140mg (N=408) | Core Phase: Oral Prophylactics (N=206) | Extension Phase: AMG334 70mg/140mg Continuing on AMG334 70mg/140mg (N=343) | Extension Phase: Oral Prophylactics Then AMG334 70mg/140mg (N=118)
Constipation (Gastrointestinal disorders) | 53 | 2 | 10 | 16
Fatigue (General disorders) | 18 | 33 | 4 | 2
COVID-19 (Infections and infestations) | 20 | 12 | 61 | 18
Nasopharyngitis (Infections and infestations) | 36 | 15 | 28 | 10
Vaccination complication (Injury, poisoning and procedural complications) | 9 | 2 | 16 | 8
Weight increased (Investigations) | 12 | 22 | 0 | 2
Dizziness (Nervous system disorders) | 7 | 18 | 6 | 1
Paraesthesia (Nervous system disorders) | 5 | 15 | 3 | 1
Somnolence (Nervous system disorders) | 5 | 15 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT03927144/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03927144/SAP_001.pdf